CLINICAL TRIAL: NCT06956976
Title: Preservation Versus Dissection of Inferior Mesenteric Artery Lymph Nodes of Robotic Radical Resection for Mid/Low Rectal Cancer (REAL2): A Multicenter Randomized Controlled Trial
Brief Title: Preservation Vs. Dissection of No. 253 Lymph Nodes of Robotic Resection for Mid/Low Rectal Cancer
Acronym: REAL2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Chair of Colorectal Surgery Department, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REAL2
Record Dates: First submitted 2025-03-25; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Rectal Cancer
Keywords: Robotic Surgery; No. 253 lymph node; lymph node dissection; disease-free survival
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IMA-LN Preservation (Active Comparator): Patients underwent robotic radical resection for rectal cancer, adhering to the principles of Total Mesorectal Excision (TME) or Tumor-Specific Mesorectal Excision (TSME), but preserving the lymph nodes at the root of the inferior mesenteric artery (IMA).
  Interventions: Procedure: Preservation of Inferior Mesenteric Artery Root Lymph Node
- IMA-LN Dissection (Placebo Comparator): Patients underwent robotic radical resection for rectal cancer, adhering to the principles of Total Mesorectal Excision (TME) or Tumor-Specific Mesorectal Excision (TSME), and dissecting the lymph nodes at the root of the inferior mesenteric artery (IMA).
  Interventions: Procedure: Dissection of Inferior Mesenteric Artery Root Lymph Node

INTERVENTIONS:
Procedure: Dissection of Inferior Mesenteric Artery Root Lymph Node — Patients underwent robotic radical resection for rectal cancer, adhering to the principles of Total Mesorectal Excision (TME) or Tumor-Specific Mesorectal Excision (TSME), and dissecting the lymph nodes at the root of the inferior mesenteric artery (IMA).
  Other Names: IMA-LN Dissection
  Arms: IMA-LN Dissection
Procedure: Preservation of Inferior Mesenteric Artery Root Lymph Node — Patients underwent robotic radical resection for rectal cancer, adhering to the principles of Total Mesorectal Excision (TME) or Tumor-Specific Mesorectal Excision (TSME), but preserving the lymph nodes at the root of the inferior mesenteric artery (IMA).
  Other Names: IMA-LN Preservation
  Arms: IMA-LN Preservation

SUMMARY:
In this study, patients with middle or low rectal cancer will receive robotic radical resection, and will be randomly assigned to receive inferior mesenteric artery lymph nodes dissection or preservation. The 3-year disease-free survival rates of these two surgical approaches will be compared.

DETAILED DESCRIPTION:
The goal of this clinical trial is to compare the outcomes of preserving versus dissecting inferior mesenteric artery root lymph nodes (IMA-LN) during robotic radical resection for mid/low rectal cancer. It aims to evaluate both short-term safety and long-term efficacy. The main questions it seeks to answer are:

1. Does preserving IMA-LN achieve non-inferior 3-year disease-free survival (DFS) compared to IMA-LN dissection?
2. Does preserving IMA-LN reduce postoperative complications (e.g., anastomotic leakage, urinary/defecation dysfunction) and improve quality of life?

Researchers will compare two surgical strategies:

1. IMA-LN preservation group: No dissection of IMA root lymph nodes, with ligation of the inferior mesenteric artery (IMA) distal to the left colic artery.
2. IMA-LN dissection group: Complete dissection of IMA root lymph nodes, with high or low ligation of the IMA.

Both groups will undergo robotic surgery following total mesorectal excision (TME) principles.

Participants will:

1. Be randomly assigned to either the preservation or dissection group. Receive standardized preoperative evaluations (imaging, biopsies) and postoperative follow-up for 3 years.
2. Undergo regular clinical assessments, including tumor marker tests, imaging (CT/MRI), colonoscopy, and quality-of-life questionnaires (evaluating urinary/sexual/defecation function).
3. Have surgical outcomes (e.g., complications, lymph node counts) and survival data recorded.

The trial aims to provide high-level evidence for optimizing surgical strategies in mid/low rectal cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years and ≤80 years
2. Pathologically confirmed rectal adenocarcinoma by colonoscopic biopsy
3. Tumor located ≤10 cm from the anal verge
4. No metastasis at the root of the inferior mesenteric artery (IMA) and no lateral lymph node metastasis confirmed by pelvic ultrasound, contrast-enhanced CT, and/or PET-CT (diagnostic criteria per the 2024 Chinese Society of Clinical Oncology [CSCO] Guidelines)
5. No distant metastasis (including pelvic, peritoneal, hepatic, pulmonary, cerebral, skeletal, or distant lymph node metastasis) confirmed by imaging
6. Pelvic MRI and/or transrectal ultrasound confirming cT1-T3 N0-1 stage, or ycT1-T3 Nx after neoadjuvant therapy (radiotherapy, chemotherapy, immunotherapy, targeted therapy)
7. No history of other malignancies (except adequately treated basal cell carcinoma or cervical carcinoma in situ)
8. Suitable for robotic surgery
9. Signed informed consent

Exclusion Criteria:

1. Clinical complete response after radiotherapy, chemotherapy, immunotherapy, or targeted therapy
2. cT1N0 tumors suitable for local excision
3. Emergency surgery required due to acute bowel obstruction, hemorrhage, or perforation
4. Multiple primary colorectal malignancies
5. Familial adenomatous polyposis (FAP), Lynch syndrome, or inflammatory bowel disease
6. Concomitant conditions requiring concurrent colonic resection
7. American Society of Anesthesiologists (ASA) grade >III
8. Pregnancy or lactation
9. Preoperative short-course radiotherapy
10. Inability of the patient/family to comprehend the study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1596 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2031-06-01 (Estimated); Study Completion 2031-06-01 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival rate | 3 years after surgery
  The 3-year disease-free survival (DFS) rate was defined as the percentage of patients with no death and no locoregional recurrence and no distant metastases within 3 years postoperatively, assessed via imaging (contrast-enhanced CT/MRI, PET-CT) or histopathological confirmation (colonoscopy/biopsy).

SECONDARY OUTCOMES:
30-day postoperative complication rate | 30 days after surgery
  The rate of patients with any of postoperative complications (Clavien-Dindo grade II or higher grade) within 30 days after surgery
Urinary function | 1 year after surgery
  Urinary function will be assessed using the International Prostate Symptom Score (IPSS) scale before surgery, at 3 months, 6 months and 1 year after surgery. For IPSS, the range of the score is 0 to 35, with higher scores indicating worse function.
Male sexual function | 1 year after surgery
  Male sexual function will be assessed using the International Index of Erectile Function-5 (IIEF-5) scale before surgery, at 3 months, 6 months and 1 year after surgery. For IIEF-5, the range of the score is 1 to 25, with lower scores indicating worse function.
Female sexual function | 1 year after surgery
  Female sexual function will be assessed using the Female Sexual Function Index (FSFI) scale before surgery, at 3 months, 6 months and 1 year after surgery. For FSFI, the range of the score is 2 to 36, with lower scores indicating worse function.
Defecation function | 1 year after surgery
  Defecation function will be assessed using the Wexner Continence Grading Scale before surgery, at 3 months, 6 months and 1 year after surgery. For the Wexner scale, the range of the score is 0 to 20, with higher scores indicating worse function.
3-year locoregional recurrence rate | 3 years after surgery
  The 3-year locoregional recurrence (LRR) rate was defined as the percentage of patients with any locoregional recurrence within 3 years postoperatively, assessed via imaging (contrast-enhanced CT/MRI, PET-CT) or histopathological confirmation (colonoscopy/biopsy).

OTHER OUTCOMES:
Intraoperative complication rate | 30 days after surgery
  Percentage of patients with any of intraoperative complications, such as: organ/structural injury (any injury requiring additional surgical repair), device malfunction (leading to procedural delay >30 minutes), fecal contamination (compromising the sterile surgical field), iatrogenic perforation (tumor or adjacent tissue perforation caused by manipulation), anastomotic complications (intraoperative anastomotic failure/leak requiring repair), tumor residual (tumor not radically resected), major hemorrhage (blood loss >200 ml at one surgical site), cardiac events (requiring intraoperative intervention), respiratory events (requiring intraoperative intervention).
Open conversion rate | 30 days after surgery
  Percentage of patients converting to open surgery.
Operative time | 30 days after surgery
  Time from skin incision to wound closure, recorded in minutes.
Estimated intraoperative blood loss | 30 days after surgery
  Calculated as suctioned blood volume + gauze weight change, recorded in ml.
Blood transfusion rate | 30 days after surgery
  Percentage of patients with any of transfusion intraoperative or within 30 days postoperatively.
Protective stoma rate | 30 days after surgery
  Percentage of patients with any of protective stoma, including terminal ileostomy or colostomy.
Macroscopic completeness of resection | 30 days after surgery
  Percentage of classification as complete, near-complete, or incomplete, according to previous report (Nagtegaal ID, et al. J Clin Oncol 2002; 20: 1729-34.)
Proximal resection margin distance | 30 days after surgery
  Distance from tumor upper edge to proximal resection margin, recorded in cm.
Distal resection margin distance | 30 days after surgery
  Distance from tumor lower edge to distal resection margin (excludes abdominoperineal resection), recorded in cm.
Distal resection margin positivity rate | 30 days after surgery
  Percentage of patients with positive distal resection margin (excluding abdominoperineal resection).
Circumferential resection margin positivity rate | 30 days after surgery
  Percentage of patients with circumferential resection margin ≤1 mm.
Number of lymph nodes harvested | 30 days after surgery
  Total number of lymph nodes detected from the specimen.
Number of No.253 lymph nodes harvested | 30 days after surgery
  Number of No. 253 lymph nodes detected at the root of inferior mesenteric artery from the specimen.
Number of positive lymph nodes | 30 days after surgery
  Number of positive lymph nodes detected from the specimen.
Number of positive No. 253 lymph nodes | 30 days after surgery
  Number of positive No. 253 lymph nodes detected at the root of inferior mesenteric artery from the specimen.
Postoperative mortality rate | 30 days after surgery
  Percentage of patients died within 30 days postoperatively.
30-day readmission rate | 30 days after surgery
  Percentage of patients with rehospitalization for disease-related causes within 30 days postoperatively.
30-day reoperation rate | 30 days after surgery
  Percentage of patients with unplanned surgery for disease-related causes within 30 days postoperatively.
Time to first flatus | 30 days after surgery
  Time from surgery completion to first passage of gas/stoma bag inflation, recorded in hour.
Time to first liquid diet | 30 days after surgery
  Time from surgery completion to first liquid intake, recorded in hour.
Time to first semi-solid diet | 30 days after surgery
  Time from surgery completion to first semi-solid intake, recorded in hour.
Time to first defecation | 30 days after surgery
  Time from surgery completion to first bowel movement, recorded in hour.
Time to first autonomous urination | 30 days after surgery
  Time from surgery completion to first autonomous urination, recorded in hour.
Postoperative hospital stay | 30 days after surgery
  Time from surgery completion to discharge, including readmissions within 30 days postoperatively, recorded in day.
3-year overall survival rate | 3 years after surgery
  The 3-year overall survival (OS) rate was defined as the percentage of patients with no death within 3 years postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Xu, Prof., Study Chair — Fudan University
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
During the recruitment process, investigators will directly contact enrolled patients to avoid privacy breaches. All identity-related data will be stored separately in locked systems and de-identified. All researchers must refrain from disclosing patients' identifiable information.
  De-identified patient data will be accessible to all investigators in this study and may be used for meta-analysis after audit and validation. Researchers should contact the principal investigator, Professor Jianmin Xu (xujmin@aliyun.com), to request data by providing a research proposal and institutional credentials. Requests will be reviewed and approved by the REAL2 trial's Independent Review Committee. Data will be available from the publication date until 36 months post-publication.
Supporting Information: Study Protocol
Time Frame: Data will be available from the publication date until 36 months post-publication.
Access Criteria: De-identified patient data will be accessible to all investigators in this study and may be used for meta-analysis after audit and validation. Researchers should contact the principal investigator, Professor Jianmin Xu (xujmin@aliyun.com), to request data by providing a research proposal and institutional credentials.